CLINICAL TRIAL: NCT00943839
Title: Effects of Sunitinib in the Expression of VEGF and of Interleukin 6 and CXCL7 - CXCL5 Cytokins : Explanation of Anti-angiogenic Effects.
Brief Title: Sunitinib Malate in Treating Patients With Kidney Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000638415; CALACASS-SUVEGIL-8; 2008/20; INCA-RECF0943; EUDRACT-2008-004137-21
Record Dates: First submitted 2009-07-21; First posted 2009-07-22 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SUVEGIL (Experimental)
  Interventions: Drug: sunitinib malate; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: sunitinib malate
Other: laboratory biomarker analysis
Other: pharmacological study

SUMMARY:
RATIONALE: Sunitinib malate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

PURPOSE: This clinical trial is studying how well sunitinib malate works in treating patients with kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine whether a link exists between the effectiveness of therapy with sunitinib malate and development of blood biomarkers, specifically the angiogenic factors VEGF and interleukin-8 (IL-8), in patients with kidney cancer.

Secondary

* To evaluate the link between the time to progression and the development of VEGF and IL-6 CXCL7 and CXCK5 blood levels in these patients.
* To evaluate the link between VEGF and IL-6 CXCL7 and CXCK5 blood levels and disease-free survival of these patients after 3, 6, 9, and 12 months of treatment.
* To evaluate the link between VEGF and IL-6 CXCL7 and CXCK5 blood levels and overall survival of these patients.

OUTLINE: This is a multicenter study.

Patients receive oral sunitinib malate once daily on days 1-28. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.

Blood samples are collected at baseline and then every 6 weeks for pharmacokinetic analysis.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed renal cell carcinoma
* Metastatic disease requiring first-line treatment with sunitinib malate

  * No prior therapy for metastatic disease
* No symptomatic or uncontrolled cerebral metastasis

PATIENT CHARACTERISTICS:

* Affiliation to the French Social insurance
* Life expectancy ≥ 3 months
* No heart failure
* No chronic unstable disease
* No long QT interval
* No history of another primary cancer
* No severe, uncontrolled acute infection
* No severe, uncontrolled hypertension
* No psychological disorder

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-02; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Disease response | 5 years
VEGF and IL-8 blood levels determined before and every 6 weeks during treatment | 5 years

SECONDARY OUTCOMES:
Length of the response | up to 5 years
Disease-free survival | up to 5 years
Overall survival | up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean Marc Ferrero, MD, Principal Investigator — Centre Antoine Lacassagne
Locations (1):
- Centre Antoine Lacassagne, Nice, France

REFERENCES:
- [Derived] Montemagno C, Durivault J, Gastaldi C, Dufies M, Vial V, He X, Ambrosetti D, Kamenskaya A, Negrier S, Bernhard JC, Borchiellini D, Cao Y, Pages G. A group of novel VEGF splice variants as alternative therapeutic targets in renal cell carcinoma. Mol Oncol. 2023 Jul;17(7):1379-1401. doi: 10.1002/1878-0261.13401. Epub 2023 Apr 18. PMID 36810959
- [Derived] Polena H, Creuzet J, Dufies M, Sidibe A, Khalil-Mgharbel A, Salomon A, Deroux A, Quesada JL, Roelants C, Filhol O, Cochet C, Blanc E, Ferlay-Segura C, Borchiellini D, Ferrero JM, Escudier B, Negrier S, Pages G, Vilgrain I. The tyrosine-kinase inhibitor sunitinib targets vascular endothelial (VE)-cadherin: a marker of response to antitumoural treatment in metastatic renal cell carcinoma. Br J Cancer. 2018 May;118(9):1179-1188. doi: 10.1038/s41416-018-0054-5. Epub 2018 Mar 22. PMID 29563634